CLINICAL TRIAL: NCT06042777
Title: Testing Non-pharmacological TCM-based Treatments for Cognitive Impairment in People With Long COVID Symptoms: A Randomized Controlled Trial
Brief Title: Non-pharmacological and TCM-based Treatment for Long COVID Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Chair Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0042751
Record Dates: First submitted 2023-09-18; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Long Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acupuncture (Experimental): This is an 8-week (two 50-min sessions per week) treatment of acupuncture on the following fixed acupoints: bilateral Touwei (ST8), Sishencong (EX-HN1), Taiyang (EX-HN5), Shuaigu (GB8), Toulinqi (GB15), and unilateral Yintang (EX-HN3), Baihui (GV20). The treatment will be performed by registered acupuncturists. based on acupuncturists' clinical judgement, acupuncture can be performed on any of the following additional acupoints, including unilateral Shenting (GV24), Shenmen (HT7), Sanyinjiao (SP6), Taichong (LV3), Neiguan (PC6), AND Anmian (EX-HN22).
  Interventions: Behavioral: Acupuncture and TCM-based lifestyle management
- TCM-based lifestyle management (Experimental): This is an integrated TCM-based training program with components of dantian breathing, Baduanjin, and self-acupressure [Yintang (EX-HN3), Shenting (GV24), Taiyang (EX-HN5), Fengchi (GB20), Neiguan (PC6), Shenmen (HT7), and Sanyinjiao (SP6)]. The treatment will last for 8 weeks (two 50-min sessions per week), and it will include health education and workshops to be delivered by trained research assistants.
  Interventions: Behavioral: Acupuncture and TCM-based lifestyle management
- Acupuncture + TCM-based lifestyle management (Experimental): This is a combination of the above two arms. The participants who randomly assigned to this arm will received two acupuncture sessions and two sessions on lifestyle management every week, and the intervention duration is 8 weeks.
  Interventions: Behavioral: Acupuncture and TCM-based lifestyle management
- Wait-list control (No Intervention): Participants will receive no intervention during the whole assessment period.

INTERVENTIONS:
Behavioral: Acupuncture and TCM-based lifestyle management — Non-pharmacological treatment based on traditional Chinese medicine.
  Arms: Acupuncture; Acupuncture + TCM-based lifestyle management; TCM-based lifestyle management

SUMMARY:
Cognitive impairment is one of the commonly reported Long COVID symptoms, mainly in terms of memory, attention, and executive function. The cognitive symptoms of Long COVID are similar to "brain fog" or "chemo brain", manifested as low energy, disorientation, difficulties in attention and communication which are common conditions in cancer patients after chemotherapy. Given the negative impact of such cognitive impairment in daily living and working, it is important to develop effective treatment and self-management techniques to enhance cognitive functions in COVID-19 survivors. Acupuncture, acupressure, dantian breathing, and qigong are promising treatment and self-management techniques to remedy the cognitive impairment in people with Long COVID. Since acupressure, dantian breathing, and qigong are feasible for self-practice, they can be trained to promote a healthy lifestyle. The present study is a randomized controlled trial to evaluate the efficacy of acupuncture, lifestyle management (including dantian breathing, qigong, and acupressure), and acupuncture + lifestyle management to improve general cognitive function of people with Long COVID symptoms, compared with wait-list control. We will recruit 100 COVID-19 survivors who experience at least mild cognitive impairment and/or self-complaint of cognitive difficulty for at least 12 weeks after clinical recovery from COVID-19 infection. They will be randomly assigned to the following groups: (1) Acupuncture Group; (2) Lifestyle Management Group; (3) Acupuncture + Lifestyle Management Group; and (4) Waitlist Control Group. Acupuncture and lifestyle management will each take 8 weeks, with two 50-min sessions per week. Primary outcome is general cognitive function. Secondary outcomes cover fatigue, physical fitness, neurocognitive function, psychological distress, and health-related quality of life, pro-inflammatory cytokines (IL-6, TNF-α) and salivary cortisol. Assessment will be conducted at baseline, mid-intervention (4 weeks after baseline), post-intervention (8 weeks after baseline), and 4-week follow-up (12 weeks after baseline).

ELIGIBILITY:
Inclusion Criteria:

* With a diagnosis of SARS-CoV-2 infection at least 3 months prior to recruitment (to be verified based on evidence of positive RT-PCR/RAT result)
* Tested negative of SARS-CoV-2 according to a RAT at the time of recruitment;
* Fulfill at least one of the following conditions: (a) With at least mild cognitive impairment as assessed with Montreal Cognitive Assessment 5-minute to be conducted by the project team; (b) Self-report of at least one cognitive symptom persisting for 12 weeks or longer after clinical recovery of SARS-CoV-2 infection according to Woods Mental Fatigue Inventory.

Exclusion Criteria:

* Having any severe cognitive impairment, mood disorder, or anxiety disorder before SARS-CoV-2 infection.
* Having any current psychiatric disorders that require taking medication.
* Having any current medical conditions that could interfere with cognitive functions.
* Having epilepsy or any other unstable medical conditions.
* Having alcoholism or drug abuse within the past 1 year.
* Having bleeding tendency.
* Having severe needle phobia.
* Having heart pacemaker or other electronic devices implanted in the body.
* Currently participating in another research studies or clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function | baseline, mid-intervention (4 weeks after baseline), post-intervention (8 weeks after baseline)
  Overall status of cognitive function

SECONDARY OUTCOMES:
Global cognitive function | baseline and 4-week follow-up (12 weeks after baseline).
  Overall status of cognitive function
Cardiopulmonary function | baseline, mid-intervention (4 weeks after baseline), post-intervention (8 weeks after baseline), and 4-week follow-up (12 weeks after baseline).
Fatigue | baseline, mid-intervention (4 weeks after baseline), post-intervention (8 weeks after baseline), and 4-week follow-up (12 weeks after baseline).
Health-related quality-of-life | baseline, mid-intervention (4 weeks after baseline), post-intervention (8 weeks after baseline), and 4-week follow-up (12 weeks after baseline).
Psychological distress | baseline, mid-intervention (4 weeks after baseline), post-intervention (8 weeks after baseline), and 4-week follow-up (12 weeks after baseline).
  Depression, anxiety, and stress
Neurocognitive functions | baseline, mid-intervention (4 weeks after baseline), post-intervention (8 weeks after baseline), and 4-week follow-up (12 weeks after baseline).
  Attention, processing speed, working memory, and executive function
Neurobiological outcomes | baseline and post-intervention (8 weeks after baseline)
  IL-6, TNF-α, and cortisol

IPD SHARING:
Plan to Share IPD: No